CLINICAL TRIAL: NCT05390879
Title: Influence of Meditation on Stress and Rumination Following Objective Structured Clinical Examination (OSCE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, Principal Investigator, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IMSR
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Stress, Psychological; Stress, Physiological; Rumination; Exam Stress
Keywords: Stress; Performance and ruminations; Coping; Rumination; Meditation; Exam; health-student
MeSH Terms: conditions — Stress, Psychological; Rumination Syndrome | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: 2 parallels groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors are blind concerning the principal outcome (ruminations and post-OSCE meditation groups, via standardized informatic questionnaires) Performance is evaluated by assessors who are blind to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Post-OSCE (Experimental): One half of the students will watch a 6 minutes auto-guided video of meditation, just after the OSCE.
  Interventions: Other: Meditation
- Control (Sham Comparator): One half of the students will watch a 6 minutes control video, just after the OSCE
  Interventions: Other: Control

INTERVENTIONS:
Other: Meditation — After the circuit, a 6 minutes long meditation auto-guided video.
  Arms: Meditation Post-OSCE
Other: Control — After the circuit, a 6 minutes long emotionally neutral video.
  Arms: Control

SUMMARY:
Stress and rumination are linked with the development of many mental disorders. The ECOSTRESS study has shown that poor OSCE performance has a positive effect on the occurence of state-rumination among 4th year medicine students in the context of mock exams.

The goal of IMSR study is to assess the effectiveness of a post-OSCE meditation intervention to decrease psychological stress and rumination.

DETAILED DESCRIPTION:
This randomized, controlled and monocentric study will be conducted during the OSCE tests contributing towards the final exam grades for 4th year medicine students at the Claude Bernard Lyon 1 university.

Before the test (OSCE), all the students will receive information about the study and formalize their consent.

The students' OSCE performance will be evaluated by an independent examiner as part of the students' exams. Upon finishing the OSCE, the students will be divided into two groups: one subjected to post-OSCE meditation and the other one subjected to a control intervention (neutral content video).

Before both interventions, all the students will be submitted to short questionnaires regarding their feelings.

During the 6-min intervention they will be get equipped with an ear pulse sensor.

Following both interventions, all the students will be submitted to short questionnaires regarding their stress and rumination levels.

The main objective is to assess the effectiveness of meditation intervention to diminish post-OSCE rumination level. The second objective is to have a deeper understanding of the cause of rumination following the OSCE..

ELIGIBILITY:
Inclusion Criteria:

* Adult person
* Registered as medical student at the university
* Participating at OSCE examination
* Have signed an informed consent form.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Change in rumination | Between before and after the intervention measured just 2 minutes before and 2 minutes after interventions (during one hour after inclusion)
  BSRI - Brief State Rumination Inventory, assessing state-rumination

SECONDARY OUTCOMES:
Physiological stress | During the 6 minutes long intervention (during one hour after inclusion)
  Heart rate variability collected by emWave® devices
Change in psychological stress level | Between before and after the intervention measured just 2 minutes before and 2 minutes after interventions (during one hour after inclusion)
  Chraracterisation of the impact of meditation on numerical Visual analog scales (VAS) on perceived stress from zero to maximum: 100mm
Change in characterisation of stress | Between before and after the intervention measured just 2 minutes before and 2 minutes after interventions (during one hour after inclusion)
  Chraracterisation of the impact of meditation on numerical VAS on characterisation of stress perceived from 0mm (negative stress) to 100mm (positive stress)
Change in self confidence | Between before and after the intervention measured just 2 minutes before and 2 minutes after interventions (during one hour after inclusion)
  Chraracterisation of the impact of meditation on numerical VAS on self confidence perceived from zero to maximum : 100mm
Rumination | One time : After intervention (during one hour after inclusion)
  Momentary Ruminative Self-focused Inventory (MRSI), 4 items long questionnaire assessing state-rumination. The goal of this outcome is to confront the french version of the MRSI (validated and published), and the newly translated BMRSI (B momentary ruminative self-focus inventory).
Feelings about the intervention | One time : After intervention (during one hour after inclusion)
  Chraracterisation of the impact of meditation on a 5 items Likert Scale (from 0: Not at all, to maximum: very high intensity) assessing feelings about the intervention: Pleasure, Interest, Enthusiasm, Boredom, Frustration, Discouragement, Fun
Change in Activation-Deactivation Adjective Check List (Thayer) | Between before and after the intervention measured just 2 minutes before and 2 minutes after interventions (during one hour after inclusion)
  Chraracterisation of the impact of meditation on activation-deactivation among students. The AD-ACL is a multidimensional test of various transitory arousal states, including energetic and tense arousal. Within the wider dimensions of energetic and tense arousal are four sub-scales-Energy (General Activation), Tiredness (Deactivation-Sleep), Tension (High Activation), and Calmness (General Deactivation), from 5 to maximum: 20 points for each dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rode, MD, PhD, Study Chair — Claude Bernard University
Locations (1):
- Marc lilot, Lyon, France